CLINICAL TRIAL: NCT01996904
Title: A Prospective Randomized Comparative Study of 191 Subscapularis Tear: Clinical and Radiologic Outcome - Arthroscopic Repair vs Debridement
Brief Title: Prospective Randomized Comparative Study of Outcome of Subscapularis Tear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CM Chungmu Hospital (Other)
Responsible Party: Principal Investigator, Sang-Hoon Lhee, Director of CM Chungmu Hospital, CM Chungmu Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CMH-2013-03
Record Dates: First submitted 2013-11-22; First posted 2013-11-27 (Estimated); Results first posted 2014-03-12 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2014-01

CONDITIONS: Rotator Cuff Syndrome
Keywords: subscapularis tear; arthroscopic tendon repair; arthroscopic tendon debridement; ASES

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- arthroscopic repair (Experimental): Lateral-anterosuperior portal ("Miracle Portal") was used to repair subscapularis tendon. Bursa anterior to the subscapularis tendon was usually removed for the accurate positioning of the suture-hook. Subscapularis tendon was released, pulled and sutured with suture-hook. One or two suture anchors of Modified Mason-Allen technique was used to secure the tendon.
  Interventions: Procedure: arthroscopic repair
- arthroscopic debridement (Active Comparator): Open and arthroscopic cuff debridement procedures have been described in the literatures for management of massive rotator cuff tears; these generally result in decreased pain and overall improvement in patient's function.
  Interventions: Procedure: arthroscopic debridement

INTERVENTIONS:
Procedure: arthroscopic repair — If the subscapularis tendon was not sufficiently mobile, further anterior interval release between subscapularis and scapula was performed. LHB (long head of biceps tendon) was either treated with a biceps tenodesis or by tenotomy when there was tear or subluxation of it. The footprint area of the subscapularis tendon, which is trapezoidal in shape on the proximal part of the lesser tuberosity, was thoroughly cleaned of soft tissue and meticulous bone preparation was done prior to placement of anchor sutures.
  Arms: arthroscopic repair
Procedure: arthroscopic debridement — Anterosuperior portal was made initially for debridement (capsulectomy and anterior bursectomy). A systematic release of the glenohumeral ligaments and the overlying subscapularis bursa was performed.The superior aspect of the tendon was freed from the surrounding structures (the coracohumeral and superior glenohumeral ligaments). The middle glenohumeral ligament was always released to identify the upper border of the subscapularis tendon.
  Arms: arthroscopic debridement

SUMMARY:
The purpose of this study was to report actual percentage of subscapularis tear in concomitant with supraspinatus tendon tear (with or without infraspinatus tear) and investigate the amount of contribution of subscapularis repair as to the outcome of whole rotator cuff repair in terms of its clinical and radiologic aspects.

DETAILED DESCRIPTION:
Prospective randomized controlled study was designed to evaluate subscapularis repair in anterosuperior rotator cuff tear compared with debridement of the subscapularis tear. After identification of the subscapularis tear arthroscopically, final eligibility of participants for the study was established on the basis of intra-operative arthroscopic inspection of the subscapularis using 70 degrees arthroscope. Once eligibility was confirmed, patients were randomized to one of two arthroscopic methods; repair (group A) or debridement (group B) of the subscapularis tear. The treatment allocations were decided through an interphone by "Research Coordinator". Block randomization was performed and no stratification was performed. Random Sequence Generator (Random.org) was used for the randomization process by given number whose digit was residue of modulo 2 (0 - group A, 1 - group B). Sequence Boundaries was 1 (smallest value) to 300 (largest value) based on the number calculated from power analysis. After randomization, patients underwent arthroscopic repair or debridement of the subscapularis tear. Size of the rotator cuff tear was also determined by the arthroscopic finding (small-to-medium, medium-to-large, large-to-massive). When full-thickness tear was confined to supraspinatus, the tear was called small-to-medium size tear. Medium-to-Large size tear was defined as complete full-thickness supraspinatus tear combined with incomplete full-thickness infraspinatus tear. Large-to-massive tear consisted of complete full-thickness tear of supraspinatus and infraspinatus or complete full-thickness tear of supraspinatus and subscapularis or complete 3-tendon tears. Postoperatively, rehabilitation was identical for both groups and consisted of sling immobilization for six weeks. Pulley exercises were performed during this time period. After six weeks from the surgery, active-assisted exercise including stick exercise to achieve full range of motion was performed. After 9 weeks from the surgery, Theraband exercise was initiated to strengthen repaired rotator cuff muscles. All patients underwent ultrasound at 24 months follow-up to evaluate integrity of supraspinatus tendon. The evaluation of integrity of supraspinatus tendon was performed and compared between two groups to evaluate the contribution of the subscapularis tendon to rotator cuff integrity. Re-tear of the supraspinatus was carefully evaluated through ultrasound by musculoskeletal radiologists who were experienced in ultrasound-diagnosis of shoulder more than 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Full-thickness supraspinatus tear confirmed by preoperative MRI
* Willingness to be enrolled into the study and understanding the whole design of the study
* Patients who is undergoing arthroscopic surgery for rotator cuff repair

Exclusion Criteria:

* An irreparable massive rotator cuff tear which shows Stage-3 or 4 fatty infiltration inside the muscle of supraspinatus and subscapularis by MRI
* Cuff tear arthropathy
* Osteoarthritis with joint space narrowing or any joint spur identified in simple radiographs
* A Workers' compensation claim
* Major trauma or rotator cuff tear after shoulder dislocation
* Previous surgery or fracture on ipsilateral extremity
* Intact subscapularis tendon identified during arthroscopic surgery with 70 degrees arthroscope

Ages: 44 Years to 83 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2009-03; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Hoon Lhee, MD, PhD, Principal Investigator — CM Chungmu Hospital
Locations (1):
- CM Chungmu Hospital, Seoul, Yeongdeungpo-gu, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: * March 2009 to October 2010
  * Out-patient department
  * Consecutive patients diagnosed with full thickness supraspinatus tear preoperative thru MRI
  * Underwent arthroscopic repair or debridement for rotator cuff tear
Pre-assignment Details: A total of 256 patients were initially identified to have subscapularis tear. They were then enrolled and all randomized. By the twenty-fourth month outcome assessment and ultrasound evaluation, 65 were lost to follow-up. 38 from group A and 27 from group B. Thus, only 191 patients making the final number of participants.
  .
Groups:
- Arthroscopic Debridement: Anterosuperior portal was made for debridement (capsulectomy and anterior bursectomy). A systematic release of the glenohumeral ligaments and the overlying subscapularis bursa was also performed. The superior aspect of the tendon was freed from the surrounding structures (the coracohumeral and superior glenohumeral ligaments). The middle glenohumeral ligament was always released to identify the upper border of the subscapularis tendon.
Period: Overall Study
Arm/Group | Arthroscopic Repair | Arthroscopic Debridement
Started | 139 | 117
Completed | 101 | 90
Not Completed | 38 | 27
Not completed — Lost to Follow-up | 38 | 27

BASELINE CHARACTERISTICS:
Population: One goal of the power analysis study design that was conducted was to test the null hypothesis, that the ASES score of two groups would be equal after undergoing treatment. The primary outcome measure was the ASES score and the secondary outcome measure includes ultrasound diagnosis until 24 months follow-up to evaluate subscapularis integrity.
Groups:
- Arthroscopic Debridement: Anterosuperior portal was made for debridement (capsulectomy and anterior bursectomy). A systematic release of the glenohumeral ligaments and the overlying subscapularis bursa was also performed. The superior aspect of the tendon was freed. from the surrounding structures (the coracohumeral and superior glenohumeral ligaments). The middle glenohumeral ligament was always released to identify the upper border of the subscapularis tendon.
- Total: Total of all reporting groups
Arm/Group | Arthroscopic Repair | Arthroscopic Debridement | Total
Number analyzed (Participants) | 101 | 90 | 191
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (5.3) | 61.6 (4.6) | 61.3 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 58 | 124
  Male | 35 | 32 | 67
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 101 | 90 | 191

OUTCOME MEASURES:

1. Primary Outcome: ASES Score
Description: The ASES is a 100-point scale which is divided in two sections. Fifty points of which are derived from patient self-report of pain and the other 50 points of which are computed from a formula using the cumulative score of 10 activities of daily living .The item related to pain is evaluated by a VAS (10 cm) that ranges from 0 (no pain at all) to 10 (pain as bad as it can be). The ten activities of daily living include skills such as putting on a coat, sleeping on the affected side, wash back/do up bra in back, manage toileting, combing one's hair, reach a high shelf, lift 10lbs above shoulder,throw a ball overhand,do usual work and do usual sport.The items related to function are evaluated by a four-point Likert scale. The scores of the pain and function subsections are transformed in percentages and each one represents 50% of the final score, which can range from 0 (absence of function) to 100 (normal function).
Time Frame: 24th month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arthroscopic Repair | Arthroscopic Debridement
Number analyzed (Participants) | 101 | 90
units on a scale | 93.3 (4.5) | 89.0 (7.3)

2. Secondary Outcome: Ultrasound Diagnosis
Description: US is a diagnostic imaging technique used to visualise deep structures of the body by recording the echoes of pulsed ultrasonic waves directed into the tissues and reflected by tissue planes to the transducer. These echoes are converted into 'pictures' of the tissues under examination. It consists of a non-invasive examination that has practically no adverse effects and allows dynamic visualisation of the tendons during movement of the shoulder.
Time Frame: every three months after the surgery until the 24th month
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Arthroscopic Repair | Arthroscopic Debridement
Serious Adverse Events (participants affected / at risk) | 0/101 | 0/90
Other Adverse Events (participants affected / at risk) | 0/101 | 0/90

LIMITATIONS AND CAVEATS:
Limitation of this study was the low retention of patients during follow-up period. Our cases only yielded 75% retention of patients after twenty-four-months follow-up and this might act as a bias in our study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No